CLINICAL TRIAL: NCT07135882
Title: A Randomised Phase III Trial of Up-front Radiotherapy Before Standard-of-care Systemic Therapy in Advanced Lung Cancer
Brief Title: Primary Radiotherapy In MEtastatic Lung Cancer
Acronym: PRIME-Lung
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Thoracic Oncology Group of Australasia (TOGA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 21.10
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung (NSCLC)
Keywords: Non-Small Cell Lung Cancer; Lung Neoplasms; Lung Cancer; Clinical reseach; Radiation Therapy; Advanced lung cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Standard of Care; Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: Standard of Care (Active Comparator): Standard of care systemic chemotherapy
  Interventions: Drug: Standard of Care (SOC)
- Arm 2: Standard of Care + Radiotherapy to primary (Active Comparator): Primary irradiation followed by standard of care systemic chemotherapy
  Interventions: Combination Product: Radiotherapy followed by chemotherapy

INTERVENTIONS:
Combination Product: Radiotherapy followed by chemotherapy — Standard of care (SoC) regimens available on the Australian PBS or relevant practice framework (Ireland and Canada) as per usual standard clinical practice are allowable in this protocol as SoC regimens.
  Radiotherapy Techniques:
  * Highly conformal techniques (IMRT/VMAT)
  * High-precision techniques are allowed for non-centrally located primaries
  Radiotherapy Dose:
  - Several fractionation schedules allowed; minimum biological effective dose approximating 50Gy (α/β ratio = 10); 50Gy in 20 fractions, 40Gy in 15 fractions, and 35Gy in 5 fractions
  Other Names: Standard of Care; Chemotherapy; Immunotherapy
  Arms: Arm 2: Standard of Care + Radiotherapy to primary
Drug: Standard of Care (SOC) — Standard of care (SoC) regimens available on the Australian PBS or relevant practice framework (Ireland and Canada) as per usual standard clinical practice are allowable in this protocol as SoC regimens.
  Other Names: chemotherapy; immunotherapy
  Arms: Arm1: Standard of Care

SUMMARY:
Lung cancer has the highest mortality rate of all cancers in Australia and is an area of unmet need. It starts in the lung (the primary tumour), and then spreads (metastasise) to other organs. The PRIME-Lung clinical trial will investigate if radiotherapy to the primary lung tumour, in addition to standard drug therapies, for patients with metastatic lung cancer will lead to less spread of cancer, prolong life, improve patient well-being and be cost-effective for the health care system.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death and is the second most common cancer in both men and women in Australia, and globally. Non-small cell lung cancer (NSCLC) accounts for 85% of cases. Almost half of the cases present with metastatic disease, in whom average survival is less than two years despite recent advances with immunotherapy. Drug therapies alone have not been able to overcome this ceiling in survival.

The primary lung tumour is a source of ongoing seeding of new metastatic (secondary) sites of disease, and we will test whether eradication of the primary tumour through non-invasive radiotherapy will limit metastases, enhance the effect of drug therapy and ultimately improve patient outcomes. Radiotherapy is a rapidly translatable solution to address this unmet need.

In the Primary Radiotherapy In MEtastatic Lung cancer (PRIME-Lung) trial, patients with metastatic NSCLC will receive standard of care systemic therapy with or without radiotherapy to the primary lung tumour. We hypothesise that radiotherapy will improve overall survival above standard of care drug therapy. PRIME-Lung is a randomised controlled phase III clinical trial and will provide a definitive answer to this critical issue.

The study team includes representation from radiation and medical oncology, physics, respiratory medicine, biostatistics, health economics and quality of life experts. The PRIME-Lung trial was designed in consultation with consumers to ensure acceptability and applicability to this area of unmet need. Furthermore, to accelerate rollout and accessibility, the trial will build on the existing AURORA lung cancer registry, leveraging the registry's established data management processes and over 25 already active sites. As radiotherapy is a pillar of oncology and widely available, upon successful completion of this trial we expect rapid translation into the community and widespread adoption of the trial results.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic (stage IV) NSCLC, not amenable to curative surgery or curative radiotherapy
* Histologically or cytologically documented NSCLC
* EGFR/ALK/ROS1 Wild-type
* Primary suitable for radiotherapy and not requiring immediate palliative thoracic irradiation
* Investigator deemed appropriate for SoC systemic therapy
* Metastases in up to 3 organ systems

Exclusion Criteria:

* Medically unfit for systemic therapy
* EGFR/ALK/ROS1 mutation positive or actionable driver mutation with intention to use available targeted drug therapy
* Has had previous thoracic radiotherapy of > 36Gy within the 6 months prior to randomisation.
* Has been diagnosed and/or treated additional malignancy within 2 years prior to randomisation with the exception of: Curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, curatively treated early-stage cervical cancer, breast cancer or prostate cancer with no evidence of active disease and not on active therapy. Other exceptions may be considered following consultation with the principal investigator
* Has a history of (non-infectious) pneumonitis or current pneumonitis that requires active corticosteroids with a dose equivalent of prednisolone > 10mg/d.
* A known diagnosis of fibrotic interstitial lung disease
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Uncontrolled brain metastasis not amenable to debulking surgery or stereotactic radiotherapy
* Has an active autoimmune disease that has required systemic treatment within last year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years after the last participant was recruited
  To assess the overall survival of patients receiving SoC systemic therapy with or without radiotherapy to the primary lung tumour

SECONDARY OUTCOMES:
Thoracic toxicity as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | 2-years after the last participant has been randomised
  To assess the safety of the addition of radiotherapy by describing thoracic toxicities of interest during the follow up period in each arm (as assessed by NCI CTCAE v5.0) and to describe the discontinuation rate of systemic therapy and reasons for discontinuation
Progression Free Survival | 2-years after the last participant has been randomised
  To assess the likelihood of progression, or death, in each arm
Cancer specific survival | 2-years after the last participant has been randomised
  To assess death from cancer-related causes in each arm
Patient Reported Quality of Life (QoL) assessed using EORTC QLQ-C30 questionnaire | 2-years after the last participant has been randomised
  To compare the effect of treatment on overall QOL, at each time point (baseline, 3, 6, 12, and 24 months) between trial arms, collected on European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Core 30 (QLQ-C30) questionnaire.
Cost effectiveness of RT plus SoC compared with SoC alone with respect to the incremental cost per quality-adjusted life year (QALYs) gained | 2-years after the last participant has been randomised
  Patient-specific costs associated with accessing care, particularly those associated with travel time for attendance, will be assessed based on questionnaires. QALYs, the combined impact of lung cancer and its treatment on survival and QoL, will be estimated by using the EORTC QLU-C10D (derived from the EORTC QLQ-C30) and EQ-5D-5L.

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, Study Chair — Peter MacCallum Cancer Centre, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Australian data will be collected using established Lung Cancer registry (AURORA). The trial sponsor is not the custodian of this registry, therefore is able to confirm IPD data can be shared at this stage.